CLINICAL TRIAL: NCT02829476
Title: Ghrelin Cellular Resistance Study in Adolescents With Idiopathic Scoliosis
Brief Title: Ghrelin Resistance in Adolescents With Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09 160 02; Local Grant 2009 (Other Grant/Funding Number: 0916002)
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Scoliosis
Keywords: Adolescent idiopathic Scoliosis; Ghrelin
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with AIS (Experimental): Patients will have 'Osteoblast sample'
  Interventions: Biological: Osteoblast sample
- control patients (Experimental)
  Interventions: Biological: Osteoblast sample

INTERVENTIONS:
Biological: Osteoblast sample — culture osteoblasts obtained from vertebrae fragments from 30 patients with AIS and from 10 control patients with secondary scoliosis

SUMMARY:
Adolescent idiopathic Scoliosis (AIS) is the most common spine pathology. It is opposed to secondary scoliosis due to chronic diseases. Many hypotheses have been made to elucidate the origin of this illness. Recently, the melatonin pathway has been investigated as pinealectomy of the chicken creates a scoliosis that resembles AIS and melatonin supplementation reverses the process. In addition administration of melatonin to AIS patients improved the pathology. However this hypothesis has shown controversial results. Recent studies have demonstrated melatonin cellular resistance in osteoblastic cells from AIS patients. Melatonin acts through G protein coupled receptor (GPCR), mainly using the Gi pathway. In AIS osteoblasts, this pathway is blocked leading to a decrease in the inactivation of the adenylyl cyclase and therefore maintenance of high level of cyclic adenosine monophosphate (cAMP) concentrations in the cells. As modulation of cAMP is important for osteogenesis such resistance may be critical for the initiation or the development of AIS.

Gi signalization is used by several other GPCR, thus, this hormonal resistance could logically be found in other hormonal or mediator pathways. A precedent study previously focused on ghrelin in AIS, and demonstrated that AIS patients possess elevated plasmatic values of ghrelin. This study also observed decreased response to ghrelin in AIS cultures osteoblasts.

ELIGIBILITY:
Inclusion Criteria:

Group 1 :

* AIS : spine deformity with angle above 10°,without detected cause
* Informed consent obtained

Group 2 :

* Secondary scoliosis due to chronic illness, neurologic or syndromic, eligible for spine surgery
* Spine surgery for reason other than scoliosis
* Informed consent obtained

Exclusion Criteria:

* Not primary scoliosis
* No consent
* Legal obstacle

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Testing ghrelin cellular resistance by intracellular cAMP dosage | baseline
  Testing ghrelin cellular resistance in AIS by measuring the variation of the intracellular cAMP level in response to ghrelin in osteoblast cells in vitro of AIS patients versus controls

SECONDARY OUTCOMES:
ghrelin level in serum | baseline
  Measure the ghrelin level in the serum of AIS patients versus controls
ghrelin levels in cellular supernatants | baseline
  Measure the ghrelin levels in cellular supernatants of osteoblasts from AIS and controls patients in order to evaluate the ghrelin production of the cells.

CONTACTS AND LOCATIONS:
Overall Officials: SALLES Jean-Pierre, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sales de Gauzy J, Gennero I, Delrous O, Salles JP, Lepage B, Accadbled F. Fasting total ghrelin levels are increased in patients with adolescent idiopathic scoliosis. Scoliosis. 2015 Nov 30;10:33. doi: 10.1186/s13013-015-0054-7. eCollection 2015. PMID 26628906